CLINICAL TRIAL: NCT07250659
Title: Comparative Effects of Intermittent Fasting Versus Mediterranean Diet on Obesity Management: A Randomized Controlled Trial
Brief Title: Comparing Intermittent Fasting and Mediterranean Diet for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kamil Dağcılar (Other)
Responsible Party: Sponsor-Investigator, Kamil Dağcılar, Assistant Professor, European University of Lefke
Organization: European University of Lefke (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAYEK011.02
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Weight Loss
Keywords: obesity; intermittent fasting; weight loss; mediterranean diet
MeSH Terms: conditions — Weight Loss; Obesity; Intermittent Fasting | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent fasting diet intervention group (Experimental): 4 week time restricted intermittent fasting diet protocol
  Interventions: Other: Intermittent Fasting Diet
- Mediterranean diet intervention group (Experimental): 4 week mediterranean diet protocol
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Intermittent Fasting Diet — Participants follow a time-restricted eating pattern for 4 weeks, consuming all meals within an 8-hour eating window (from 1:00 PM to 9:00 PM) and fasting for the remaining 16 hours each day. During the feeding window, they consume two main meals and one snack based on ad libitum intake, without specific calorie restriction. Dietary guidance is provided at the start and mid-point of the protocol by a registered dietitian.
  Arms: intermittent fasting diet intervention group
Other: Mediterranean Diet — Participants follow a 4-week Mediterranean diet protocol that is adapted from the PREDIMED criteria and the MedDietScore index. The diet emphasizes high consumption of vegetables, fruits, legumes, whole grains, nuts, and olive oil; moderate intake of fish and poultry; and limited consumption of red meat, dairy products, and sweets. A registered dietitian provides dietary counseling sessions at the beginning and midway through the intervention.
  Arms: Mediterranean diet intervention group

SUMMARY:
Purpose: This study aimed to evaluate and compare the effects of intermittent fasting (IF) and the Mediterranean diet (MD) on weight loss in obese adults.

Methods: A total of 120 adults diagnosed with obesity were enrolled. Baseline data on physical activity and dietary intake were collected through structured interviews. Participants were randomly assigned to two groups for a 4-week intervention. The IF group followed a time-restricted eating schedule (16:8), while the MD group followed a structured plan of three main meals and three snacks daily. Both diets included a 500-calorie daily reduction from estimated energy needs. Anthropometric measurements were recorded at baseline and week 4.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m²
* absence of chronic diseases
* no regular use of medications
* non smokers
* non alcohol users
* not pregnant or breastfeeding
* no history of bariatric surgery
* no significant weight fluctuations (±5 kg) in the past 6 months
* no pregnancy plans during the study period

Exclusion Criteria:

* BMI < 30 kg/m²
* Presence of any diagnosed chronic disease (e.g., diabetes, cardiovascular disease, thyroid disorders, renal or hepatic disease)
* Regular use of medications that could affect metabolism, appetite, or body weight
* Smoking or alcohol consumption
* Pregnancy or breastfeeding during the study period
* History of bariatric or other weight-related surgical procedures
* Significant weight changes (gain or loss ≥5 kg) within the past 6 months
* Planning pregnancy during the study period
* Inability or unwillingness to comply with dietary intervention and follow-up requirements

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) | Baseline and Week 4
  Body weight is measured with using the TANITA BC-418 body composition analyzer. Participants are weighed barefoot, in light clothing, and measurements are recorded in kilograms.

SECONDARY OUTCOMES:
Body Mass Index (kg/m²) | Baseline and Week 4
  BMI is computed as weight in kilograms divided by height in meters squared (kg/m²)

OTHER OUTCOMES:
Body height (cm) | Baseline only
  Height is measured once at baseline using a wall-mounted stadiometer. Participants stand barefoot, with heels together, arms at the sides, and head positioned in the Frankfurt horizontal plane. The measurement is recorded to the nearest 0.1 centimeter and converted to meters.
Body Fat Percentage | Baseline and week 4
  Body fat percentage is measured at baseline and Week 4 using the TANITA BC-418 body composition analyzer
Fat Free Mass (kg) | Baseline and Week 4
  Fat free mass is assessed using bioelectrical impedance analysis with TANITA BC-418
Total Body Water Percentage | Baseline and Week 4
  Total body water percentage is assessed using bioelectrical impedance analysis with TANITA BC-418.
Waist Circumference (cm) | Baseline and Week 4
  Waist circumference is measured using a non-elastic, flexible measuring tape. The measurement is taken at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest, while the participant stands upright with feet close together and breathes out normally.
Hip Circumference (cm) | Baseline and Week 4
  Hip circumference is measured with using a non-elastic measuring tape. The measurement is taken around the widest portion of the buttocks, with the participant standing upright and feet together.

CONTACTS AND LOCATIONS:
Locations (1):
- European University of Lefke, Lefka, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (1):
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT07250659/ICF_000.pdf